CLINICAL TRIAL: NCT04181957
Title: The Effects of Lisdexamfetamine Dimesylate on Cognitive, Metabolic, and Reward Processes in Individuals With Binge-eating Symptoms
Brief Title: Effects of LDX on Cognitive Processes and Appetite
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRAS 250510
Record Dates: First submitted 2019-11-13; First posted 2019-12-02 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2019-01

CONDITIONS: Binge Eating; Eating Behavior
MeSH Terms: conditions — Bulimia; Feeding Behavior | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Intervention Model Description: Counter-balanced, double-blind, placebo-controlled, crossover, within-subject design.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The research is double-blind. The pharmacists have prepared active and placebo capsules of LDX identical in appearance, and a scientist on the project who is not associated with data collection randomises the condition based on a random, counter-balanced design. The resulting capsule's contents are blind to the participant, data collectors, and the prescribing physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants receive placebo tablet composed of lactose.
  Interventions: Drug: Placebo oral tablet
- Active (Active Comparator): Participants receive a 50mg tablet of lisdexamfetamine dimesylate (LDX) once.
  Interventions: Drug: Lisdexamfetamine Dimesylate

INTERVENTIONS:
Drug: Placebo oral tablet — Participants take one dose of placebo (lactose) tablet.
  Arms: Placebo
Drug: Lisdexamfetamine Dimesylate — Participants take one 50mg tablet of lisdexamfetamine dimesylate once.
  Arms: Active

SUMMARY:
This study will investigate the effect of lisdexamfetamine dimesylate (LDX) on the mediating factors of reward and cognition on appetite.

DETAILED DESCRIPTION:
This study will investigate the specific reward and cognitive mechanisms that mediate the effects of LDX on eating in participants with sub-clinical binge-eating disorder symptoms. A sub-clinical sample will be recruited in line with the Research Domain Criteria Initiative established by the US National Institute of Mental Health which encourages research on dimensions of observable behaviour rather than a categorical, symptom-based approach to the study of mental health. The tendency towards binge-like eating will be modelled using an eating in the absence of hunger paradigm in which participants consume a pasta meal and are then offered the opportunity to consume as many palatable cookies as they like. Reward processes will be assessed by measuring neural and behavioural responses to palatable food pictures using functional Magnetic Resonance Imaging (fMRI). Responses to emotional stimuli will be assessed using the P1vital® Oxford Emotional Test Battery. Impulsive responding will be assessed using the delay discounting task and the stop signal task. Attentional processing will be assessed using the sustained performance task and working memory will be assessed with the n-back task.

ELIGIBILITY:
Inclusion Criteria:

* Fluent English speakers
* Be willing to be informed of chance pathological findings from the fMRI scan
* Must have binge-eating symptoms that is measured by a minimum score of 18 on the Binge Eating Scale
* Must have a minimum BMI of 18.5
* Must be below 152.4kg
* Must have clearance from a qualified physician before participating

Exclusion Criteria:

* Symptoms or diagnosis of other eating disorders.

  * Psychotherapy and/or pharmacotherapy for binge-eating disorder (BED) 3 months before the study, as this will suggest a diagnosis of BED and may influence eating behaviour.
  * Metabolic (e.g. metabolic disorder, diabetes), psychological (e.g. depression), substance, or neurological (e.g. epilepsy, headache disorder, multiple sclerosis, traumatic brain injuries) diseases or medication in relation to these diseases
  * Intake of any medication that can interfere with the drug or measurements, determined through questionnaires in the screening session
  * Current smoking, as it can interfere with appetite
  * Current pregnancy or breastfeeding
  * Not passing a breathalyser test on the morning of testing.
  * Food allergies (e.g. peanut allergy, lactose and gluten intolerance) or vegetarian/vegan diet
  * Disliking the study lunch to ensure that participants will consume the provided food
  * Women will be asked to participate only in weeks when they are not menstruating or in their pre-menstrual week, to avoid hormonal disruption to appetite.

The following are exclusion criteria are specific to the MRI scanner:

* Non-removable metal object in or on their body, such as: heart pace-maker, artificial heart valve, metal prosthesis, implants or splinters, non-removable dental braces
* Left-handed
* Tattoos that are older than 10 years
* Claustrophobia
* Limited temperature perception and/or increased sensitivity to warming of the body
* Pathological hearing ability or an increased sensitivity to loud noises
* Operation less than three months ago
* Simultaneous participation in other studies that involve drug intake or blood sampling
* Acute illness or infection during the last 4 weeks
* Cardiovascular disorders (e.g., hypertrophic cardiomyopathy, long QT syndrome) to ensure medical fitness to participate
* Moderate or severe head injury

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Metabolic food intake | 15 minutes
  We will examine if LDX has an influence on metabolic food intake using a lab-based food task, in which participants eat as much pasta as they like until they feel comfortably full . Amount eaten will be measured in grams.
Hedonic food intake | 15 minutes
  The effect of LDX on hedonic food intake will be measured via offering a palatable snack of chocolate chip cookies 20 minutes after participants have consumed the pasta. Amount eaten will be measured in grams.

SECONDARY OUTCOMES:
fMRI Reward Processes | 21 minutes
  We will investigate the effect of LDX on neural responses to food stimuli using fMRI, and if/how liking ratings modulate these responses. The participants will perform a food and non-food rating task in the scanner, to measure reward-responses. Participants will view a range (36 each category) of high -and low-calorie food (equally distributed in sweet and savoury), and non-food items (visually matched). All items will be scored for appealing/liking with the use of a button box, varying from 1 (not at all) to 5 (very much). Each item will be presented for 3000ms followed by a fixation cross (500 - 1500ms). (3 x 7 min = 21 min)
Ratings | 20 minutes
  We will determine if LDX administration has an effect on appetite and mood ratings via a visual analogue scale (VAS) in a hungry and sated state. Participants will drag a cursor from 0cm (not at all) to 10cm (most I could imagine) to self-report mood and appetite.
Emotional processing | 35 minutes
  We will determine if LDX modulates emotional processing. The ETB is a computerised battery that comprises the following tasks:
  FERT: Faces will appear on a screen ranging in emotions. The participant is instructed to classify each expression as quickly and accurately as possible. Accuracy, response bias, reaction time, and target sensitivity.
  ECAT: 60 positive and negative adjectives will be presented for the participant to indicate if they would like to be described as such. Accuracy and reaction times.
  EREC: The participants will be asked to recall as many words from the ECAT as can be remembered within a 4-minute period. The number of correct words recalled and respective valence will be measured.
  EMEM: Participants will be presented with personality descriptors derived from the ECAT, along with matching novel distractor words. Participants will indicate if the descriptor was presented before. Accuracy, reaction time, response bias, and target sensitivity.
Memory | 10 minutes
  We will investigate the effect of LDX on working memory. To assess working memory and working memory capacity, participants will complete a visuospatial n-back task. The participant is presented with a sequence of circles on a 3x3 grid. The participant is instructed to indicate whether the current circle location matches the location of the circle n trials earlier. In this design, participants will identify if the circle matches the circle 2 and 3 trials back on separate cycles. Participants will complete 70 trials of each n-back condition. This task takes approximately 10 minutes to complete.
Attention | 14 minutes
  We will investigate the effect of LDX on attention. This task is a series of white letters presented on a grey background in random order, modelled on the Conner's Continuous Performance Task. Participants are instructed to press the space bar for every letter except 'X'. Letters will be presented for 900ms. Accuracy and reaction time will be measured. The task duration is 14 minutes.
Cognitive inhibition/Impulsivity | 10 minutes
  We will investigate LDX effect on cognitive control (ie inhibition). Participants will complete the delay-discounting task for money and food. The delay-discounting task measures the extent to which participants are willing to delay the receipt of a reward, in exchange for receiving a higher-value reward, and is generally considered to reflect impulsive behaviour. This task is a monetary discounting task with nine delays ranging from one day to one year. On a screen, participants see the question 'Which would you prefer?', with two choices: £xx now or £xx after a delay (varying from one day to one year), and will be asked to choose between the two. A similar paradigm will be used for food, with questions consisting of food variables instead of money. Questions will require a choice between a smaller amount of food now, and a larger amount later. Area under the curve will be calculated.
Motor inhibition/Impulsivity | 10 minutes
  We will measure the effect of LDX on inhibition using the Stop Signal Task. The stop signal task requires the participant to identify the direction of a circle's location on the screen (i.e., left or right). If, however, the circle is encased in another circle, then the participant is to withhold a response. Successful inhibition, commission errors, and reaction time will be measured.
fMRI food reward - activation | 21 minutes
  We will investigate the activation changes in brain regions associated with reward to food when viewing pictures of food.
  When assessing changes in activation we will assess how activity in separate brain regions changes when attending to food pictures compared to when attending to visually-matched non-food pictures.
fMRI food reward - functional connectivity | 21 minutes
  We will investigate the changes in functional connectivity between brain regions associated with reward to food when viewing pictures of food.
  When looking at changes in functional connectivity we will assess how the relationship between activity in any two or more brain regions is altered when attending to food pictures compared to when attending to visually-matched non-food pictures.
fMRI inhibition - activation | 18 minutes
  We will investigate the effect of LDX on brain regions associated with cognitive control, during performance of a delay discounting task (Outcome 8). When assessing changes in activation we will assess how activity in separate brain regions changes when making decisions about food compared to when making decisions about money.
fMRI inhibition - functional connectivity | 18 minutes
  We will investigate the changes in functional connectivity between brain regions associated with cognitive control.
  When looking at changes in functional connectivity we will assess how the relationship between activity in any two or more brain regions is altered when making decisions about food compared to when making decisions about money.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Higgs, PhD, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Open access to study protocol and data.
Supporting Information: Study Protocol
Time Frame: The study protocol and data will become available after the last participant has finished the study.
Access Criteria: All researchers